CLINICAL TRIAL: NCT03663296
Title: Assessing Usefulness of Virtual Reality Mobile Application in Flexible Videoscope Airway Training - a Randomised Controlled Trial
Brief Title: Assessing Usefulness of Virtual Reality Mobile Application in Flexible Videoscope Airway Training
Acronym: AURA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AURA
Record Dates: First submitted 2018-09-02; First posted 2018-09-10 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Education, Medical

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Additional 30 minutes of self-directed learning and practice using the mobile application, after conventional training session
  Interventions: Other: Airway Ex App
- Control (No Intervention): Conventional training session which includes didactic teaching and low-fidelity simulation session involving trainer's demonstration, followed by hands-on practice

INTERVENTIONS:
Other: Airway Ex App — 30 minutes of self-directed learning and practice using the mobile application
  Arms: Interventional

SUMMARY:
Flexible videoscope orotracheal intubation (FOI) technique is considered an important option in the management of predicted difficult airways. However, it is rarely performed in daily practice. Yet emergency physicians are expected to be able to perform this skill expertly during a crisis scenario. If it is not completed in a timely and proper fashion, the patient will deteriorate rapidly, resulting in morbidity or fatality.

There is a significant learning curve to master this complex psychomotor skill. Providing sufficient training in FOI, particularly hands-on experience in real patients is difficult. Patients with known difficult airway requiring FOI present infrequently to the emergency room. Using patients with normal airway purely for teaching of FOI is ethically controversial. To avoid technical and ethical concerns of training involving real patients, conventional teaching methods incorporate the use of a low-fidelity manikin in replacement. However, the manikin anatomy often lacks the realism of a live human.

The addition of virtual reality technology, in the form of a low-cost mobile application (Airway Ex) into the conventional simulation, may optimize learning by providing an ethical, cost-effective and more realistic modality to acquire the basic skills of FOI. If it is proven to be effective, efforts to integrate virtual reality technology into routine training of such procedures in the ED should be promoted.

We hypothesize that the addition of virtual reality mobile application to conventional training will improve procedural skill dexterity and proficiency and hence, improve learner's satisfaction and confidence in performing FOI.

ELIGIBILITY:
Inclusion Criteria:

* All doctors from Accidental & Emergency Department of National University Hospital, Singapore

Exclusion Criteria:

* Refusal for consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2018-08-11 (Actual); Study Completion 2019-08-11 (Actual)

PRIMARY OUTCOMES:
Time taken for successful intubation | 5 minutes
  time from advancing scope from manikin's mouth to confirmed placement of endotracheal tube through visualisation with videoscope

SECONDARY OUTCOMES:
Time taken for visualisation of vocal cords | 1 minute
  time from advancing scope from manikin's mouth to first visualisation of vocal cords with videoscope

OTHER OUTCOMES:
Quality of flexible videoscope manipulation ability | 5 minutes
  By blinded assessor using validated Five-point Global Rating Scale of Fiberoptic Bronchoscope Manipulation Ability. Score of 1 indicates very poor techniques whereas a score of 5 indicates clearly superior techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Wei Yau, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No